CLINICAL TRIAL: NCT01212458
Title: Effect of Oral Rufinamide and Oxcarbazepine on Nerve Excitability, Hyperalgesia, Allodynia and Flare Reaction Compared to Placebo. A Monocenter, Randomized, Double-blind, Cross-over Study
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Version 1.03
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Subjects
Keywords: gesunde Probanden

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Rufinamid — Effect of oral rufinamide and oxcarbazepine on nerve excitability, hyperalgesia, allodynia and flare reaction compared to placebo.

SUMMARY:
Untersuchungen über die Wirkmechanismen von Antiepileptika haben gezeigt, dass durch eine Blockierung von spannungsabhängigen Natrium-Kanälen im Nervensystem die Schmerzübertragung moduliert werden kann. Verschiedene Antiepileptika werden in der chronischen Schmerztherapie schon lange angewendet (z.B. Oxcarbazepinum, Trileptal ® bei Trigeminusneuralgie oder diabetischer Polyneuropathie).

In unserer Untersuchung wollen wir zwei in der Schweiz zugelassene Antiepileptika bezüglich ihrer Wirkung auf das Schmerzempfinden untersuchen. Eines dieser Medikamente, Trileptal® (Wirkstoff: Oxcarbazepinum), wird schon häufig bei chronischen Schmerzzuständen eingesetzt. Das zweite Medikament, Inovelon® (Wirkstoff: Rufinamid) ist seit mehr als einem Jahr in der Schweiz zugelassen und wird klinisch vor allem in der Behandlung von besonderen Epilepsieformen im Kindesalter eingesetzt. Wir erwarten, dass auch nach Gabe von Inovelon® die Schmerzleitung in den Nervenzellen verändert und die lokalen Schmerzreaktionen in der Haut vermindert werden.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria: Male

* Age: 18-65 years
* Weight: 50 - 100 kg
* Height: 155 - 195 cm
* Signed and dated informed consent

Exclusion criteria:

* Contraindications to the class of drugs under study
* Intellectually or mental impaired subjects
* Known hypersensitivity to class of drugs or the investigational product
* Drug abuse
* Known peripheral neuropathies
* Diabetes mellitus
* Chronic alcohol consumption
* Congestive heart disease
* Participants of other studies during study period and 30 days prior to study begin
* Smoker
* Abnormal electrocardiogram
* Any regular concomitant medication

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Maurer, MD, Principal Investigator — University Hospital Zurich, Institut of Anaesthesiology
Locations (1):
- University Hospital Zurich, Institut of Anaesthesiology, Zurich, Canton of Zurich, Switzerland